CLINICAL TRIAL: NCT01210378
Title: Nitroglycerin as a Sensitizer in the Treatment of Non Small Cell Lung Cancer: a Phase II Trial
Brief Title: Nitroglycerin in Non-small Cell Lung Cancer
Acronym: Nitroglycerin
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Accrual stopped
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Reliable Cancer Therapies (Industry); Anticancer Fund, Belgium (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nitroglycerin in NSCLC
Record Dates: First submitted 2010-09-27; First posted 2010-09-28 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Non Small Cell Lung Cancer (NSCLC)
Keywords: NSCLC; Nitroglycerin; Tumour perfusion; Hypoxia; Toxicity; Phase II; HX4
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Hypoxia | interventions — Nitroglycerin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nitroglycerin (Experimental)
  Interventions: Drug: Nitroglycerin patch

INTERVENTIONS:
Drug: Nitroglycerin patch — Nitroglycerin patch

SUMMARY:
Nitroglycerin is a nitric oxide donor which is mainly known as a vasodilating agent used in ischemic heart disease. It has also been shown to increase tumor blood flow in animal and human tumors.

The addition of nitroglycerin to chemotherapy in non small cell lung cancer has been shown to generate very favorable response rates with respect to standard treatment schedules[5]. Theoretically nitroglycerin might reduce resistance to chemotherapy via a plethora of different effects: better tumor perfusion, direct effects of NO on cancer cells, increase in activated p53 protein and via an increased blood flow in the tumour with as consequence a higher drug concentration in the tumor [6] .

In mice, nitric oxide donors such as isosorbide dinitrate have been shown to decrease tumor hypoxia by better tumor perfusion, which could enhance radiotherapy responses [7].

To date these combined effects have not been tested in humans. In this trial we would like to demonstrate the effect of nitroglycerin on tumor perfusion and hypoxia in non small cell lung cancer (using DCE and HX4 scanning), providing a rationale for further study and to test the effect of combining nitroglycerine to standard treatment of NSCLC (radiotherapy/chemotherapy).

DETAILED DESCRIPTION:
Namely, the failure of many different tumor types to show a lasting response chemotherapy or radiotherapy might be attributable to a lack of oxygen supply (called "hypoxia" from hereon) in a large part of the cancer cells.

Tumor hypoxia is a well-known factor negatively influencing outcome in many solid tumors, including lung cancer, head and neck cancer, etc. Hypoxic cells are more radio-resistant, more chemo-resistant and more prone to develop distant metastases than normoxic cells.

Nitroglycerin, due to it's vasoactive effects, tends to redistribute the blood supply to the tumor, increasing tumor blood flow, hereby theoretically decreasing hypoxia.

It has been shown that NO donating drugs can alter tumor blood flow and oxygenation status in animal models [7]. In a randomized phase 2 trial by Yasuda nitroglycerin has been successfully combined at a dose of 25 mg daily for 5 days each chemo cycle with cisplatin and vinorelbine in non small cell lung cancer, enhancing chemotherapy response, possibly due to better delivery of the anti-cancer drugs in the tumor[5]. The toxicity profile between the 2 arms was not significantly different.

The effects of nitroglycerin or other donating drugs on cancer have been found to be numerous: not only is there an increase in tumor bloodflow, also direct effects on stabilization of p53 and degradation of Hif-1 alpha have been found[6]. Decreased hypoxic biomarkers (eg VEGF, P-glycoprotein) have been found in patients with NSCLC treated with nitroglycerin patches for 3 days prior to surgery when compared to non-treated individuals [8]. There might also be a supplementary effect on the MHC-molecules, rendering tumor cells more "visible" to the immune system [9].

Furthermore, hypoxia has been shown in vitro to increase the invasiveness of cancer cells in an NO-mediated manner, which can be blocked by NO-donors.[10] An interesting study in this respect is a non-randomized phase 2 trial by Siemens et al, in which a very low dose of nitroglycerin (Minitran 5 patch (18 mg) cut in 6 pieces, delivering 0.033 mg/h in stead of 0.2 mg/h normally) was given to patients with biochemical recurrence (PSA-failure) after primary therapy. After 24 months the PSA doubling time was more than 31 months versus 12.8 months before the start of therapy, demonstrating the inhibitory effect of nitroglycerin on prostate cancer cells. [11]

Due to these effects and the effect on tumor bloodflow and decrease of hypoxia nitroglycerin might also be interesting as a radiosensitizing agent.

Currently a Mexican phase 2 trial is recruiting 40 patients to evaluate the efficacy of nitroglycerin added to concurrent chemoradiotherapy in NSCLC stage III. (Clinical trials.gov identifier NCT00886405).

The aim of the present study is not only to demonstrate the effect of nitroglycerin on perfusion and hypoxia through (HX4-)scanning of patients, but also documenting the efficacy of the approach of giving nitroglycerin in an on/off (12h/12h) schedule to people receiving (chemo-)/radiotherapy, whilst monitoring toxicity.

The on-off schedule is chosen because of the existence of a tolerance effect on the vascular system, hence diminishing the effect of nitroglycerin already after the first 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Non-small cell lung cancer stage IB-IV amenable for radiotherapy with curative intent.
* (Stage IV patients with oligometastic (1-4 metastases) NSCLC are regularly treated radically in the IKNL region).
* Patients not included in the PET-Boost or the Lucanix trial.
* WHO performance status 0-2.
* Willing and able to comply with the study prescriptions.
* 18 years or older.
* Ability to give and having given written informed consent before patient registration.
* No recent (< 3 months) severe cardiac disease (NYHA class >1) (congestive heart failure, infarction).
* No radiotherapy in 4 weeks prior to this study.
* No treatment with investigational drugs in 4 weeks prior to or during this study.
* No known allergy to nitroglycerin or nitroglycerin patch.
* No known allergy to iodine based contrast agents
* No use of Levitra, Viagra or Cialis at the time of application of the nitroglycerin patch.
* No conditions necessitating the use of ergot alkaloids, alpha blockers (eg tamsulosine), betablockers or calcium channel blockers on the day of nitroglycerin patch application).
* No other active malignancy.
* No major surgery (excluding diagnostic procedures like eg mediastinoscopy) in previous 4 weeks.
* Adequate renal function: calculated creatinine clearance at least 60ml/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Increase of 2 year overall survival of 15% vs historical controls | 2 years

SECONDARY OUTCOMES:
Demonstrate effect on enhancement on tumor perfusion | 3 days
Toxicity | 7 weeks
Demonstrate the effect on enhancement of tumor oxygenation | 3 days
Evaluating the possible value of Perfusion CT and hypoxia scans on treatment with nitroglycerin of NSCLC | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lambin, MD, PhD, Principal Investigator — Maastro Clinic, The Netherlands
Locations (1):
- MAASTRO clinic, Maastricht, Netherlands

REFERENCES:
- [Derived] van Elmpt W, Zegers CML, Reymen B, Even AJG, Dingemans AC, Oellers M, Wildberger JE, Mottaghy FM, Das M, Troost EGC, Lambin P. Multiparametric imaging of patient and tumour heterogeneity in non-small-cell lung cancer: quantification of tumour hypoxia, metabolism and perfusion. Eur J Nucl Med Mol Imaging. 2016 Feb;43(2):240-248. doi: 10.1007/s00259-015-3169-4. Epub 2015 Sep 4. PMID 26338178